CLINICAL TRIAL: NCT05091164
Title: Feasibility Study of Sleep Endoscopy Under Hypnosis in a Sleep Center
Acronym: DISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: European Clinical Trial Experts Network (Other); Polyclinique Poitiers (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-A02419-30
Record Dates: First submitted 2021-10-15; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Drug Induce Sleep Endoscopy; Hypnosis; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate obstructive sleep apnea syndrome patient under hypnosis (Experimental): Patients suffering from moderate obstructive sleep apnea syndrome. It is proposed to induce in the patient a hypnotic trance leading to intense muscle relaxation, capable of reproducing in the upper airways.
  The type of collapsibility thus obtained, classified according to Kezirian (6), will allow specific management by OAM in the event of predominant anteroposterior stenosis.
  Interventions: Procedure: Drug induce sleep endoscopy of upper aerodigestive tract under hypnosis

INTERVENTIONS:
Procedure: Drug induce sleep endoscopy of upper aerodigestive tract under hypnosis — Drug induce sleep endoscopy of upper aerodigestive tract under hypnosis.

SUMMARY:
It is proposed to induce in a obstructive sleep apnea syndrome patient, a hypnotic trance leading to intense muscle relaxation, capable of reproducing in the upper airways (VAS) the muscle relaxation observed in sleep, at the origin of obstructive apnea and snoring. The collapsibility type obtained, classified according to Kezirian, will allow specific management by OAM in the event of predominant anteroposterior stenosis. There are no risks fort the patient. The Drug Induce Sleep endoscopy (DISE) is a fibroscopy of upper aerodigestive tract.

ELIGIBILITY:
Inclusion Criteria:

* Patient, women or men over 18 years old
* Moderate obstructive sleep apnea syndrome (Hypopnea apnea index between 15 and 30) without any serious sign
* Simple Ronchopathy
* Indication of video-fibroscopy of upper airways
* Affiliated subject or beneficiary of a social security scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Psychiatric disorders that can be decompensated by hypnosis (bipolarity, schizophrenia, ...)
* Smoking less than 10 cigarettes per day
* Alcoholism, chronic or serious disabling pathology
* Medical history of cancer of upper airways, radiotherapy
* Pregnancy
* Recent supper airway infection, rhinosinusitis
* Active allergy
* Non-obstructive sleep apnea syndrome
* severe non-obstructive sleep apnea syndrome (Hypopnea apnea index> 30)
* Dental contraindication to mandibular advancement device
* Intolerance or allergy to local anesthesia with Xylocaine spray 5% known
* Refusal to participate in the study
* Protected patients: adults under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant, breastfeeding or parturient woman
* Hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-04-08 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
proportion of patients for whom the DISE could be performed in good conditions of comfort | 45 days
  The good conditions of comfort for the patient, the operator and the healthcare professional trained in hypnosis will be evaluated using a comfort scale with 4 subscales of 5 items, rated from 1 to 4, in Likert scale from 1 (not at all satisfied) to 4 (very satisfied), i.e. for each subscale a sub-score between 5 and 20 and an overall score between 20 and 80.
  * Patient comfort
    * Physical comfort (5 items)
    * Psychological comfort (5 items)
  * Practitioner comfort
    o For the realization of the DISE (5 items)
  * Comfort of the health professional trained in hypnosis o For the realization of hypnosis (5 items) It will be considered that the DISE could have been carried out in good conditions of comfort (for the patient, the operator and the healthcare professional trained in hypnosis), if the overall score is ≥60 AND no sub-score n 'is <10.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre du Sommeil de la Polyclinique de Poitiers, Potiers, France